CLINICAL TRIAL: NCT03881267
Title: A Multi-center, Randomized Controlled Clinical Trial Evaluating the Effects of SkinTE® in the Treatment of Venous Leg Ulcers
Brief Title: SkinTE® in the Treatment of Venous Leg Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PolarityTE (Industry)
Collaborators: Professional Education and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STE-VLU-01
Record Dates: First submitted 2019-03-17; First posted 2019-03-19 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Venous Leg Ulcer; Venous Stasis; Venous Stasis Ulcer
Keywords: VLU; Ulcer; SkinTE
MeSH Terms: conditions — Varicose Ulcer; Ulcer

STUDY DESIGN:
Intervention Model Description: Multi-center, Randomized Controlled Clinical Trial Evaluating the Effect of Human Homologous Autologous Skin Construct (SkinTE™) in the Treatment of Venous Leg Ulcers
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human Autologous Homologous Skin Construct (SkinTE) (Experimental): SkinTE, is an autologous, homologous, FDA-registered, cutaneous human cellular and tissue-based product (HCT/P) that can be used an adjunct to standard of care, for skin coverage in patients who have suffered from a venous leg wound in conjunction with standard wound care and Additional (outer) Dressing Application with moisture retention dressing and compression
  Interventions: Other: Human Autologous Homologous Skin Construct; Other: Additional Outer Dressing Application
- Fibracol Wound Dressing (Active Comparator): A commercially available wound dressing to be used per manufacturer's instructions for use on venous leg wounds in conjunction with standard wound care and Additional (outer) Dressing Application with moisture retention dressing moisture retention dressing and compression
  Interventions: Other: Additional Outer Dressing Application; Other: Fibracol Wound Dressing

INTERVENTIONS:
Other: Human Autologous Homologous Skin Construct — Application of a autologous human derived skin polar units
  Other Names: SkinTE
  Arms: Human Autologous Homologous Skin Construct (SkinTE)
Other: Additional Outer Dressing Application — Application of Moisture retentive dressing, and a multi-layer compression dressing
  Other Names: •Outer protective and compressive dressing
Other: Fibracol Wound Dressing — Application of Collagen Alginate Dressing
  Other Names: Collegen Alginate
  Arms: Fibracol Wound Dressing

SUMMARY:
This study is a prospective, multi-center, randomized controlled trial designed to collect patient outcome data on a commercially available human autologous homologous skin construct with SOC dressing compared to SOC dressings alone in the treatment of Venous Leg Wounds

DETAILED DESCRIPTION:
This study is a prospective, multi-center, Randomized Controlled Trial (RCT) designed to collect patient outcome data on a commercially available human autologous homologous skin construct (SkinTE) with SOC dressing compared to SOC dressings alone in the treatment of Venous Leg Wounds (VLU). The trial will be single blinded in regard to wound healing assessment (another clinician, other than the investigator at each site will assess wound healing) and confirmation of wound healing will be overseen by an independent adjudication committee made up of wound care experts. The study will last twelve weeks, with a two week screening period prior to enrollment.

There are two arms in the study:

Arm 1: The Experimental Arm , that will include SOC Therapy. SOC therapy in this study is appropriate sharp or surgical debridement, infection management (systemic antibiotics only in conjunction with debridement) and the experimental wound care covering with human autologous,homologous skin construct (SkinTE) followed by a moisture retention dressing and a padded 3-layer dressing comprised of 4x4 gauze pads, soft roll and compression wrap (DynaflexTM or equivalent).

Arm 2: The Standard of Care Arm. The SOC therapy in this study is appropriate sharp or surgical debridement, infection management (systemic antibiotics only in conjunction with debridement) and wound care covering with calcium alginate Fibracol dressing followed by a moisture retentive dressing and a padded 3-layer dressing comprised of 4x4 gauze pads, soft roll and compressive wrap (DynaflexTM or equivalent).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Presence of a VLU on the leg, below the knee but above the aspect of the medial malleolus, extending at least through the dermis or subcutaneous tissue but not involving tendon, muscle, or bone.
* The index ulcer will be the largest ulcer if two or more VLUs are present and will be the only one evaluated in the study. If other ulcerations are present on the same foot, they must be more than 2 cm distant from the index ulcer.
* Index ulcer (i.e. current episode of ulceration) has been present for greater than four weeks prior to the initial screening visit, as of the date subject consents for study.
* Index ulcer is a minimum of 2.0 cm2 and a maximum of 20 cm2 at first screening visit (SV1) and first treatment visit (TV1).
* Adequate circulation to the affected extremity as documented by a dorsal transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg, or an Ankle Branchial Index (ABI) between ≥ 0.7 and ≤ 1.2 or Arterial Doppler with a minimum of biphasic flow within 3 months of SV1, using the affected study extremity.
* The index ulcer has been treated with high compression for at least 14 days prior to randomization (30-40 mm Hg).
* Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers or abstinence) during the course of the study and undergo pregnancy tests.
* Subject understands and is willing to participate in the clinical study and can comply with weekly visits and follow-up regimen.
* Subject has read and signed the IRB/IEC approved Informed Consent Form before screening procedures have been completed.
* The index ulcer has a clean granular base, is free of necrotic debris, and appears to be healthy vascularized tissue at time of placement of treatment product.
* Subject is deemed healthy and stable for treatment based per PI discretion.

Exclusion Criteria:

* Subjects with a BMI ≥45
* Index ulcer(s) deemed by the investigator to be caused by a medical condition other than venous insufficiency.
* Known allergy to the components of the multi-layer compression bandaging, or who cannot tolerate multi-layer compression therapy.
* Index ulcer, in the opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a carcinoma of the ulcer.
* Subjects on any investigational drug(s) or therapeutic device(s) within 30 days preceding the first Screening Visit (SV1).
* History of radiation at the ulcer site (regardless of time since last radiation treatment).
* Index ulcer has been previously treated or will need to be treated with any prohibited therapies, such as chlorhexidine or collagenase. (See Section 7.3 of this protocol for a list of prohibited medications and therapies).
* Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids > 10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to first Screening visit, or who receive such medications during the screening period, or who are anticipated to require such medications during the study.
* Study ulcer requiring negative pressure wound therapy during the course of the trial.
* Ulcers on the dorsum of the foot or with more than 50% of the ulcer below the malleolus are excluded.
* Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence with medical treatment.
* Subject is pregnant or breast-feeding.
* Presence of diabetes with poor metabolic control as documented with an HbA1c ≥12.0 within 30 days of randomization.
* Subjects with end stage renal disease as evidenced by a creatinine greater than 3.0mg/dl within 120 days of randomization.
* Target wound has presence of local active soft tissue infection involving the treatment site.
* Index ulcer has reduced in area by 30% or more after 14 days of SOC from SV1 to the TV1/randomization visit.
* In the opinion of the Investigator, evidence of unstable human immunodeficiency virus (HIV), hepatitis B or hepatitis C at screening.
* Vascular surgery; arterial or venous to the affected extremity within 30 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Percentage of index ulcers healed at 12 weeks | 12 weeks
  examine percent of ulcers healed at week twelve

SECONDARY OUTCOMES:
Percentage area reduction at 4 weeks | 4 weeks
  examine percent of wound reduction at 4 weeks
Percentage area reduction at 6 weeks | 6 weeks
  examine percent of wound reduction at 6 weeks
Percentage area reduction at 8 weeks | 8 weeks
  examine percent of wound reduction at 8 weeks
Percentage are reduction at 12 weeks | 12 weeks
  examine percent of wound reduction at 12 weeks
Improvement in quality of life using Wound Quality of Life Score | 12 weeks
  The Wound-QoL, or wound quality of life questionnaire, measures the disease-specific, health-related quality of life of patients with chronic wounds. It consists of 17 items on impairments which are always assessed in retrospect to the preceding seven days. This questionnaire will be given to clinical trial participants at each visit, with the scale scores recorded. Each question is scored. Answers to each item are coded with numbers (0='not at all' to 4='very much'). As noted above the score will be reported with a minimam score of "0" and a maximum score of 68
Change in pain levels during trial, using the FACES pain scales which measure pain on a range of 0-10, zero being no pain and 10 being the most severe pain | 12 weeks
  The FACES pain scale will be administered to the clinical trial participants at each visit. The trial participant will select their pain level with a series of faces that correspond to a number between 0 which implies no pain , up to 10 which implies the most severe pain. The scores will be recorded for each clinical trial participant on each visit

OTHER OUTCOMES:
Visible Graft Take at each visit | 12 weeks
  Examine the take or the bodies ability to accept the Skin TE

CONTACTS AND LOCATIONS:
Overall Officials: David Armstrong, DPM, MD, PhD, Principal Investigator — USC/ Salsa
Locations (2):
- United States (2):
  - Martinsville Research Institute, Martinsville, Virginia
  - Professional Education and Research Institute, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No